CLINICAL TRIAL: NCT02742818
Title: Forced-air Warming in Endovascular Surgery: Testing Effectiveness of Two Different Blanket Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nelson Wolosker (Other)
Responsible Party: Sponsor-Investigator, Nelson Wolosker, MD, PHD, Hospital Israelita Albert Einstein
Organization: Hospital Israelita Albert Einstein (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Forced-air warming in ES
Record Dates: First submitted 2016-03-30; First posted 2016-04-19 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Hypothermia
Keywords: forced-air warming; hypothermia; endovascular surgery; blanket
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Upper body blanket, Bair Hugger (Other): Patients undergoing EVAR and LEA will use this type of warming blanket.
  Interventions: Device: Upper body blanket, Bair Hugger
- Underbody blanket, Bair Hugger (Other): Patients undergoing EVAR and LEA will use this type of warming blanket.
  Interventions: Device: Underbody blanket, Bair Hugger

INTERVENTIONS:
Device: Upper body blanket, Bair Hugger — Upper body warming blanket will be used in patients undergoing LEA and EVAR.
  Arms: Upper body blanket, Bair Hugger
Device: Underbody blanket, Bair Hugger — Underbody warming blanket will be used in patients undergoing LEA and EVAR.
  Arms: Underbody blanket, Bair Hugger

SUMMARY:
Prospective randomized trial comparing effectiveness of two different forced-air warming blankets in patients undergoing lower extremity angioplasty (LEA) and endovascular abdominal aortic aneurysm repair (EVAR).

DETAILED DESCRIPTION:
Fifty patients undergoing LEA and EVAR will be randomized into two groups: Group upper body blanket and Group underbody blanket. All patients will receive general anesthesia and body temperature will be measured and registered by an esophageal thermometer with 15 minutes interval beginning immediately after tracheal intubation up to tracheal extubation. The warming unit used (Bair Hugger 750 warming unit, Arizant Healthcare) will be the same for both groups and the blankets tested will be: upper body blanket (Bair Hugger 522 upper body blanket, 3M) and underbody blanket (Bair Hugger 635 full acess underbody blanket, 3M). Surgical and anesthetic complications will be noted. Only surgeries with minimum 45 minutes duration will be accepted for the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing LEA and EVAR
* American Society of Anesthesiologists physical status (ASA) : 1-4

Exclusion Criteria:

* Non-endovascular surgery
* pregnant patients
* patient refusal
* less than 45 minutes duration of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Upper Body Blanket: Patients undergoing EVAR and LEA will use this type of warming blanket.
  522 upper body blanket, Bair Hugger, 3M
- Underbody Blanket: Patients undergoing EVAR and LEA will use this type of warming blanket.
  635 full access underbody blanket, Bair Hugger, 3M
Period: Overall Study
Arm/Group | Upper Body Blanket | Underbody Blanket
Started | 25 | 25
Completed | 25 | 23
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Underbody Blanket | Upper Body Blanket | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [60.5 to 76.5] | 70 [62 to 73] | 70.5 [60.25 to 74.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 15 | 19 | 34

OUTCOME MEASURES:

1. Primary Outcome: Values of Body Temperature ( in Celsius Degree ) in Two Groups of Patients Undergoing EVAR and LEA That Will Use Two Different Types of Bair Hugger 3M Body Warming Blankets, Namely: 522 Upper Body Blanket and 635 Full Access Underbody Blanket.
Description: After tracheal intubation, upper body or underbody blanket will be turned on at the highest temperature of the warming unit ( 43 celsius degree) and the body temperatures will be measured and registered with an esophageal thermometer every 15 minutes until tracheal extubation. Temperatures will be compared with the purposes of determining which one of the two models tested are more effective in keeping patient warm. Values of body temperature across duration of surgery will be compared by models of variance analysis with repeated measurements. Duration of surgery will be used as a control variable.
Time Frame: Across duration of surgery (up to 210 minutes)
Population: In the Underbody blanket group 2 patients were excluded from analysis. One of the patients due to anaphylactic reaction and the other framed exclusion criteria (Surgery time lesser than 45 minutes)
Measure: Median (Full Range); unit: Celsius degrees
Arm/Group | Upper Body Blanket | Underbody Blanket
Number analyzed (Participants) | 25 | 23
Celsius degrees | 36.2 [35.1 to 37.3] | 36.1 [34.3 to 37.1]
Statistical Analysis 1: Comparison: Upper Body Blanket vs Underbody Blanket; Test type: Other; p = 0.190, Generalized Estimation Equations (GEE); Model assuming Gaussian distribution and AR-1 correlation structure, considering repeated measures in time; Through inference, changes in body temperature and proportional occurrence of hypothermia during surgery were evaluated using general models of estimating equations (GEE, Liang e Zeger, 1986). Binominal and normal distributions were taken into account, respectively, and assumptions for errors normalities were verified using residual plot graphs and fitted values. The significance of other associated factors and probable outcomes were verified, including gender, age, surgery type and total surgery duration, in minutes. Since analyses were longitudinal, AR-1 working correlation matrix was created

2. Secondary Outcome: Age ( in Years)
Description: The investigators will observe the profile of the patients and the mean of age in two groups.
Time Frame: At time of surgery ( in minutes)
Measure: Median (Inter-Quartile Range); unit: years
Arm/Group | Upper Body Blanket | Underbody Blanket
Number analyzed (Participants) | 25 | 23
years | 70 [62 to 73] | 71 [60.5 to 76.5]
Statistical Analysis 1: Comparison: Upper Body Blanket vs Underbody Blanket; Test type: Other; p = 0.820, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Gender
Description: The investigators will observe gender distribution in the two groups studied.
Time Frame: At time of surgery ( in minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Underbody Blanket | Upper Body Blanket
Number analyzed (Participants) | 23 | 25
Participants
  Male | 15 | 19
  Female | 8 | 6
Statistical Analysis 1: Comparison: Underbody Blanket vs Upper Body Blanket; Test type: Other; p = 0.529, Chi-squared

4. Secondary Outcome: Type of Surgery ( LEA and EVAR )
Description: The investigators will observe the type of surgery distribution profile in the two groups studied.
Time Frame: At time of surgery ( in minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Upper Body Blanket | Underbody Blanket
Number analyzed (Participants) | 25 | 23
Participants
  EVAR | 13 | 12
  LEA | 12 | 11
Statistical Analysis 1: Comparison: Upper Body Blanket vs Underbody Blanket; Test type: Other; p = 0.999, Chi-squared

5. Secondary Outcome: Duration of Surgery ( in Minutes)
Description: The investigators will observe the duration of surgery (in minutes) in the two groups studied.
Time Frame: Across duration of surgery ( in minutes)
Population: Models of generalized estimation equations will be used to evaluate the evolution of body temperature across duration of surgery (in minutes)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Upper Body Blanket | Underbody Blanket
Number analyzed (Participants) | 25 | 23
minutes | 180 [150 to 210] | 210 [135 to 232.5]
Statistical Analysis 1: Comparison: Upper Body Blanket vs Underbody Blanket; Test type: Other; p = 0.462, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Upper Body Blanket | Underbody Blanket
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 0/25 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upper Body Blanket (N=25) | Underbody Blanket (N=25)
Anaphylatic reaction (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Upper Body Blanket (N=25) | Underbody Blanket (N=25)
Anaphylatic reaction (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No